CLINICAL TRIAL: NCT07237347
Title: Perceptions and Ultrasound Literacy for Sound Volume Management
Acronym: PULSE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: am25Loosen;Req-2025-00684
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ultrasound-guided Fluid Management; Volume Responsiveness; Venous Congestion Assessment; ICU Physician Practices
Keywords: Ultrasound; fluid management; volume responsiveness; intensive care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU staff: physicians working in ICUs in Switzerland
  Interventions: Other: Quastionnaire

INTERVENTIONS:
Other: Quastionnaire — physicians working in ICUs will complete a questionnaire through REDcap

SUMMARY:
The aim of this study is to assess the knowledge, attitudes, and practices of ICU physicians in Switzerland regarding the use of ultrasound for fluid management and evaluation of venous congestion.

DETAILED DESCRIPTION:
This multicenter survey study aims to explore the experiences, perceptions, and attitudes of intensive care unit (ICU) physicians in Switzerland regarding the use of ultrasound for fluid management. The primary objective is to assess participants' knowledge of ultrasound techniques to predict fluid responsiveness and evaluate venous congestion. The study will also compare familiarity with traditional methods (e.g., central venous pressure, IVC-Inferior Vena Cava ultrasound) and newer approaches such as the VEXUS (Venous Excess Ultrasound Score) score or assessment of stroke volume changes during passive leg raise or mini fluid challenges.

Participants will complete an online questionnaire via REDCap, covering demographics, professional background, ultrasound training, knowledge and experience with ultrasound for volume management and venous congestion, as well as institutional factors and suggestions for improvement. The survey will be distributed to physicians working in ICUs at multiple Swiss hospitals, including the University Hospital Basel, Kantonsspital Aarau, Inselspital Bern, Spitalzentrum Biel, and Triemlispital Zürich. Participation is voluntary, and informed consent will be obtained electronically at the start of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* physicians working in ICUs
* working in Switzerland

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: physicians working in Swiss ICUs
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Physician Knowledge and Experience Using Ultrasound for Fluid Management and Venous Congestion | completion of questionnaire takes about 30 minutes
  The primary outcome is the proportion of ICU physicians in Switzerland who demonstrate knowledge and report regular use of ultrasound techniques for assessing fluid responsiveness and venous congestion, including traditional methods and newer approaches. Data will be collected through a structured online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Loosen, MD, Principal Investigator — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No